CLINICAL TRIAL: NCT05428306
Title: Pharmacokinetic Interaction Study Between Ibuprofen 200 mg and Acetaminophen 500 mg, Tablets Administered Individually or in Combination, Single Dose in Healthy Subjects, Both Genders Under Fasting Conditions
Brief Title: Pharmacokinetic Interaction Between Ibuprofen and Acetaminophen, Tablets Administered Individually or in Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BD IP-Sil No.103-18
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Pharmacokinetic; No interaction; Fixed-dose combination (FDC); Ibuprofen; Acetaminophen; Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Ibuprofen/ Acetaminophen in fixed dose (Experimental): Pharmaceutical Form: Tablet Formula: Ibuprofen 200 mg/ Acetaminophen 500 mg Dosage: 400 mg / 1000 mg (2 tablets) Administration way: oral
  Interventions: Drug: A1: Ibuprofen/Acetaminophen Fixed dose combination (Laboratorios Silanes S.A. de C.V.)
- Group B: Ibuprofen (Active Comparator): Pharmaceutical Form: tablets Dosage: 400 mg (1 tablet) Administration way: oral
  Interventions: Drug: A2: Ibuprofen (Motrin®, Pfizer S.A. de C.V.)
- Group C: Acetaminophen (Active Comparator): Pharmaceutical Form: Tablet Formula: Acetaminophen 500 mg Dosage: 1000 mg (2 tablets) Administration way: oral
  Interventions: Drug: A3: Acetaminophen (Tylenol caplets®, from Janssen-Cilag, S.A. de C.V.)

INTERVENTIONS:
Drug: A1: Ibuprofen/Acetaminophen Fixed dose combination (Laboratorios Silanes S.A. de C.V.) — Formula : 200 mg/ 500 mg Pharmaceutical Form: Tablet Dosage: 400 mg / 1000 mg (2 tablets) Administration way: oral
  Other Names: IBU / ACETA
  Arms: Group A: Ibuprofen/ Acetaminophen in fixed dose
Drug: A2: Ibuprofen (Motrin®, Pfizer S.A. de C.V.) — A2: Pharmaceutical Form: tablet Dosage: 400 mg (1 tablet) Administration way: oral
  Other Names: IBU
  Arms: Group B: Ibuprofen
Drug: A3: Acetaminophen (Tylenol caplets®, from Janssen-Cilag, S.A. de C.V.) — A3:Pharmaceutical Form: tablet Formula: Acetaminophen 500 mg Dosage: 1000 mg (2 tablets) Administration way: oral
  Other Names: ACETA
  Arms: Group C: Acetaminophen

SUMMARY:
This study was carried out in the Clinical and Analytical Unit of the Pharmacology and Toxicology Department of the Faculty of Medicine of the Autonomous University of Nuevo León, with the aim of comparing the bioavailability (Cmax, AUC) of an oral formulation containing ibuprofen 400 mg/ Acetaminophen 1000 mg in combination with the two oral formulations ibuprofen 400 mg or Acetaminophen 1000 mg administered as a single dose, in healthy subjects under fasting conditions

DETAILED DESCRIPTION:
The study design was crossover, 3 x 6 x 3, open, prospective and longitudinal, at a single dose of the combination of Ibuprofen 200mg/ Acetaminophen 500mg (2 tablets), administered orally versus each component administered individually Ibuprofen 400mg (1 tablet) or Acetaminophen 500 mg (2 tablets), with three treatments, three periods, six sequences with an elimination period (washout) of 1 week and with a number of 42 healthy subjects, of both genders, under fasting conditions. In order to compare the pharmacokinetic profile (Cmax and AUC 0-t) of the combination Ibuporfen/Acetaminophen 200 mg / 500 mg, single dose versus each component administered individually, to establish the non-interaction of the drugs in combination. Like, Characterize the pharmacokinetic parameters, Cmax and AUC 0-t, AUC 0-, Tmax, Ke and T1/2, of Ibuprofen and Acetaminophen after oral administration in a single dose. The frequency and type of adverse events with the two formulations were established.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must have been accepted by the COFEPRIS research subjects registration database.
* Subjects without a subordinate relationship with the researchers.
* Subjects who have given informed consent in writing.
* Subjects of both genders, aged between 18 and 55 years, Mexicans.
* Subjects with no background of hypersensitivity or allergies to the drug under study or related drugs.
* Body mass index between 18 and 27 kg/m2.
* Healthy subjects, according to the results of the complete clinical history, electrocardiogram and the integration of the results of the clinical analyses, carried out in certified clinical laboratories, without alterations that require a medical intervention as a consequence.
* Subjects with negative results for immunological tests (Anti-HIV, Anti-hepatitis B and C, VDRL).
* Subjects with negative results in drug abuse screening tests: tetrahydrocannabinoids, cocaine and amphetamines.
* Negative (qualitative) pregnancy test for women of childbearing potential without Bilateral tubal obstruction or hysterectomy.
* In the case of women of childbearing age, they must have a birth control method, including barrier methods, non-hormonal intrauterine device, or bilateral tubal obstruction.

Exclusion Criteria:

* Subjects with recent history or physical examination evidence of gastrointestinal, renal, hepatic, endocrine, respiratory, cardiovascular, dermatological, or hematological disease that could affect the pharmacokinetic study of the product in research.
* Subjects who have been exposed to drugs known as liver enzyme inducers or inhibitors or who have taken drugs potentially toxic within 30 days before the start of the study.
* Subjects who have received any medication during the 7 days before the start of the study.
* Subjects who have been hospitalized for any problem during the three months before the start of the study.
* Subjects who have been rejected by the registry database of research subjects of COFEPRIS, for having participated in a clinical study within the three months prior to the start of the study.
* Subjects who have received investigational drugs within the previous 60 days th the start of the study.
* Subjects allergic to the study drug or related drugs.
* Subjects who have ingested alcohol or drinks containing xanthines (coffee, tea, cocoa, chocolate, cola) or who have eaten charcoal-grilled food or grapefruit juice , at least 10 hours before the start of the study or who have smoked tobacco 24 hours before to the start of the internment period.
* Subjects who have donated or lost 450 mL or more of blood within the previous 60 days of the beginning of the study.
* Subjects with a history of drug and/or alcohol abuse according to the DSM-IV-TR Criteria.
* Research subjects who presents alterations in the vital signs recorded during the selection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration following the treatment (Cmax), | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours
  Evaluate the pharmacokinetics profile of the fixed dose Ibuprofen/Acetaminophen, employing the maximum observed concentration following the treatment (Cmax), obtained graphically, from the plasma concentration profile with respect to time.
The area under the curve from time zero to the last measurable concentration (AUC 0-t) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours
  Evaluate the fixed dose pharmacokinetics profile of Ibuprofen/Acetaminophen, employing the area under the curve from time zero to the last measurable concentration (AUC 0-t) using the linear trapezoidal method.

SECONDARY OUTCOMES:
The area under the curve from time zero to infinity calculated (AUC 0-inf) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours
  Evaluate the fixed dose pharmacokinetics profile of Ibuprofen/Acetaminophen, employing the area under the curve from time zero to infinity calculated (AUC 0-inf).
Time of the maximum measured concentration (Tmax) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours
  Evaluate the fixed dose pharmacokinetics profile of Ibuprofen/Acetaminophen employing time of the maximum measured concentration Tmax), Obtained graphically, from the plasma concentration profile with respect to time.
Elimination rate (Ke) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours
  Evaluate the fixed dose pharmacokinetics profile of Ibuprofen/Acetaminophen, employing the elimination rate (Ke), estimated from the terminal linear portion of the plasma concentration profile with respect to time (on a semi-log scale)
Half time elimination (t1/2) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours
  Evaluate the pharmacokinetics profile of the fixed dose Ibuprofen/Acetaminophen, employing the half time elimination (t1/2) by the quotient of Ln(2)Ke.
Frequency of occurrence of adverse events | 1, 8 and 16 days
  The percentage of frequency of appearance of each adverse event was evaluated.
Adverse Events | 1, 8 and 16 days
  Any adverse event were classified by severity, treatment and its relationship with the study drug was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Garza Ocaña, M.D, Principal Investigator — Department of Pharmacology and Toxicology of the Faculty of Medicine of the U.A.N.L
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson BJ. Paracetamol (Acetaminophen): mechanisms of action. Paediatr Anaesth. 2008 Oct;18(10):915-21. doi: 10.1111/j.1460-9592.2008.02764.x. PMID 18811827
- [Background] Bramlage P, Goldis A. Bioequivalence study of three ibuprofen formulations after single dose administration in healthy volunteers. BMC Pharmacol. 2008 Oct 29;8:18. doi: 10.1186/1471-2210-8-18. PMID 18959779
- [Background] Tanner T, Aspley S, Munn A, Thomas T. The pharmacokinetic profile of a novel fixed-dose combination tablet of ibuprofen and paracetamol. BMC Clin Pharmacol. 2010 Jul 5;10:10. doi: 10.1186/1472-6904-10-10. PMID 20602760
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848